CLINICAL TRIAL: NCT00042198
Title: Treatment of Depression After Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kenneth Freedland, Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH060735 (NIH); R01MH060735 (NIH); DSIR AT-AS
Record Dates: First submitted 2002-07-24; First posted 2002-07-26 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Depression; Coronary Disease
Keywords: Cognitive therapy; Relaxation techniques
MeSH Terms: conditions — Depression; Coronary Disease | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Cognitive Behavior Therapy. The treatment modality was individual, face-to-face therapy with an experienced cognitive therapist. Treatment consisted of up to 12 weekly, hour-long sessions.
  Interventions: Behavioral: Cognitive behavior therapy
- 2 (Active Comparator): Supportive Stress Management. The treatment modality was individual, face-to-face therapy with an experienced psychotherapist. Treatment consisted of up to 12 weekly, hour-long sessions.
  Interventions: Behavioral: Supportive Stress Management
- 3 (No Intervention): Usual Care, minimally enhanced. Participants in all three arms were given information about depression. There were no restrictions in any of the arms on usual care for depression, heart disease, or any other conditions, except that concurrent participation in nonstudy psychotherapy was not allowed. Participants were allowed to continue or start on nonstudy antidepressants during the study, as prescribed by the participant's personal physician.

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — Up to 12 weekly, individual, hour-long sessions
  Arms: 1
Behavioral: Supportive Stress Management — Up to 12 weekly, individual, hour-long sessions, focusing on application of relaxation and other stress management techniques to depressogenic stressors
  Arms: 2

SUMMARY:
This randomized controlled trial will test the efficacy of (1) cognitive behavior therapy and (2) supportive stress management as treatments for depression in people who have recently undergone coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
Depression is a very common problem for people who have had CABG surgery, and recent studies have shown that it may increase the risk of additional medical problems and death during the first few years after surgery. Cognitive behavior therapy (CBT) has been shown to be efficacious for depression in otherwise healthy individuals, and supportive stress management (SSM) interventions have also been shown to improve depressive symptoms. These therapies have not, however, been tested for depression in individuals who have undergone CABG surgery.

Participants will be screened for depression within 1 year after CABG surgery. Those who have depression will return for additional testing 1 week later. Eligible participants will be randomized to receive CBT, SSM, or usual care (UC), with no restrictions on nonstudy antidepressants, for 12 weeks. Patients will be monitored for worsening depression referred for additional care if needed. Depression, anxiety, and health-related quality of life will be assessed at baseline, 12 weeks after randomization, and 6 months after surgery (2 months after termination of CBT or SSM).

ELIGIBILITY:
Inclusion Criteria:

* Coronary Artery Bypass Graft (CABG) surgery (alone or combined with valvular or carotid surgery) within past 12 months
* Meets DSM-IV criteria for major or minor depressive episode

Exclusion Criteria:

* Severe cognitive impairment
* Severe psychiatric comorbidity (e.g., alcoholism or schizophrenia)
* Severely debilitating or life-threatening illness other than coronary disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2001-12; Primary Completion 2005-12 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D-17) | 12 weeks post-randomization
  The HAM-D-17 is an observer-rated measure of the severity of depression.

SECONDARY OUTCOMES:
Beck Depression Inventory | 12 weeks post-randomization
  The BDI is a self-report measure of the severity of depression.
Beck Anxiety Inventory | 12 weeks post-randomization
  The BAI is a self-report measure of the severity of anxiety symptoms.
Beck Hopelessness Scale | 12 weeks post-randomization
  The BHS is a self-report measure of hopelessness.
Perceived Stress Scale | 12 weeks post-randomization
  The PSS is a self-report measure of perceived stress
SF-36 | 12 weeks post-randomization
  The Medical Outcomes Study SF-36 is a measure of health-related quality of life. The Physical and Mental factor scores will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E Freedland, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Freedland KE, Skala JA, Carney RM, Rubin EH, Lustman PJ, Davila-Roman VG, Steinmeyer BC, Hogue CW Jr. Treatment of depression after coronary artery bypass surgery: a randomized controlled trial. Arch Gen Psychiatry. 2009 Apr;66(4):387-96. doi: 10.1001/archgenpsychiatry.2009.7. PMID 19349308
- See also: Volunteer for Health--Washington University's research volunteer program — http://vfh.wustl.edu/